CLINICAL TRIAL: NCT01034852
Title: Surgery After Previous Failed Catheter Ablation
Brief Title: Efficacy Study for Surgery After Previous Failed Catheter Ablation
Acronym: SAVED
Status: Completed | Type: Observational
Sponsor: Cardiopulmonary Research Science and Technology Institute (Other)
Collaborators: AtriCure, Inc. (Industry); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.018
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Atrial Fibrillation Ablation
Keywords: Atrial Fibrillation; Maze; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — no biospecimens will be obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical ablation: Patients undergoing surgical ablation for Atrial Fibrillation that have failed one or more previous attempts at catheter ablation for Atrial Fibrillation
  Interventions: Procedure: Totally Thoracoscopic Maze

INTERVENTIONS:
Procedure: Totally Thoracoscopic Maze — Epicardial pulmonary vein isolation with additional lesions as determined to be necessary by physician
  Other Names: Minimally invasive maze; Cox Maze procedure

SUMMARY:
Specific Aims: The primary objective of this registry is to determine the percentage of patients who are free from atrial fibrillation (AF) at 6 and 12 months following a surgical ablation procedure when the patient has a history of failing one or more previous catheter based ablations for AF. The first 3 months following surgical ablation will be a blanking period; any arrhythmia occurring during this time will not be used to determine success.

Primary Objectives:

1. Determine the percent success of surgical ablation for AF at 6, and 12 months both on and off of antiarrhythmic drugs (AAD) following a failed catheter based ablation for AF
2. Record and evaluate all complications associated with the surgical procedure.

Secondary Objectives:

1. Evaluate usage of anticoagulants at 6, and 12 months.
2. Determine the percentage of Pulmonary Veins (PV) that were electrically isolated by intra-operative, pre-surgical mapping

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atrial fibrillation
* Has undergone one or more catheter based ablation procedures for AF and the procedure failed
* Has undergone a minimal access surgical ablation procedure for the treatment of AF following failure of catheter based ablation for AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone surgical ablation after failing catheter based ablation at investigator sites
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of surgical ablation for AF at 6, & 12 months both on and off of antiarrhythmic drugs following a failed catheter based ablation for AF. | 1 year post operatively
Record and evaluate all complications associated with the surgical procedure. | 1 year post operatively

SECONDARY OUTCOMES:
Evaluate usage of anticoagulants at 6 and 12 months. | 1 year post operatively
Determine the % of Pulmonary Veins that were electrically isolated by intra-operative, pre-surgical mapping. | 1 year post operatively

CONTACTS AND LOCATIONS:
Overall Officials: James R Edgerton, MD, Principal Investigator — Cardiopulmonary Research Science and Technology Institute
Locations (2):
- United States (2):
  - Endovascular Research, Springfield, Oregon
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas